CLINICAL TRIAL: NCT03194620
Title: Absorption, Metabolism and Excretion of Dietary Polyphenolic Bioactives in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 907244
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Flavanols; Cocoa Flavanols; Epicatechins; Polyphenols; Procyanidins; EGCG; EGC; ECG; Theaflavins; Thearubigins
MeSH Terms: interventions — theaflavin; epigallocatechin gallate; epicatechin gallate; Catechin; gallocatechol

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked and cross-over dietary intervention study in healthy young adult males
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control (Placebo Comparator): Single oral intake of flavanol-free fruit-flavored non-dairy drink
  Interventions: Other: Control
- Theaflavins (Experimental): Single oral intake of a fruit-flavored non-dairy drink containing a mixture of theaflavins
  Interventions: Other: Theaflavins
- Procyanidin Dimer B2 (DB2) (Experimental): Single oral intake of a fruit-flavored non-dairy drink containing Procyanidin Dimer B2 (DB2)
  Interventions: Other: Procyanidin Dimer B2 (DB2)
- (-)-Epigallocatechin-3-O-gallate (EGCG) (Experimental): Single oral intake of a fruit-flavored non-dairy drink containing (-)-Epigallocatechin-3-O-gallate (EGCG)
  Interventions: Other: (-)-Epigallocatechin-3-O-gallate (EGCG)
- (-)-Epicatechin-3-O-gallate (ECG) (Experimental): Single oral intake of a fruit-flavored non-dairy drink containing (-)-Epicatechin-3-O-gallate (ECG)
  Interventions: Other: (-)-Epicatechin-3-O-gallate (ECG)
- (-)-Epicatechin (EC) (Active Comparator): Single oral intake of a fruit-flavored non-dairy drink containing (-)-Epicatechin (EC)
  Interventions: Other: (-)-Epicatechin (EC)
- (-)-Epigallocatechin (EGC) (Experimental): Single oral intake of a fruit-flavored non-dairy drink containing (-)-Epigallocatechin (EGC)
  Interventions: Other: (-)-Epigallocatechin (EGC)
- Thearubigins (Experimental): Single oral intake of a fruit-flavored non-dairy drink containing thearubigins
  Interventions: Other: Thearubigins

INTERVENTIONS:
Other: Thearubigins — Single oral intake of 94.9 mg of therubigins (isolated from black tea) in a flavanol-free, fruit flavored, non-dairy drink
  Arms: Thearubigins
Other: Theaflavins — Single oral intake of 120 µmol of an equimolar mixture of theaflavins (isolated from black tea) in a flavanol-free, fruit flavored, non-dairy drink. The theaflavin mix includes theaflavin, theaflavin-3-gallate and theaflavin-3,3'-gallate
  Arms: Theaflavins
Other: Procyanidin Dimer B2 (DB2) — Single oral intake of 120 µmol of Procyanidin Dimer B2 (DB2) (isolated from Theobroma cacao) in a flavanol-free, fruit flavored, non-dairy drink.
  Arms: Procyanidin Dimer B2 (DB2)
Other: (-)-Epigallocatechin-3-O-gallate (EGCG) — Single oral intake of 120 µmol of (-)-Epigallocatechin-3-O-gallate (EGCG)(isolated from green tea) in a flavanol-free, fruit flavored, non-dairy drink.
  Arms: (-)-Epigallocatechin-3-O-gallate (EGCG)
Other: (-)-Epicatechin-3-O-gallate (ECG) — Single oral intake of 120 µmol of (-)-Epicatechin-3-O-gallate (ECG) (isolated from green tea) in a flavanol-free, fruit flavored, non-dairy drink.
  Arms: (-)-Epicatechin-3-O-gallate (ECG)
Other: (-)-Epicatechin (EC) — Single oral intake of 120 µmol of (-)-Epicatechin (EC) (isolated from green tea) in a flavanol-free, fruit flavored, non-dairy drink.
  Arms: (-)-Epicatechin (EC)
Other: (-)-Epigallocatechin (EGC) — Single oral intake of 120 µmol of (-)-Epigallocatechin (EGC) (isolated from green tea) in a flavanol-free, fruit flavored, non-dairy drink.
  Arms: (-)-Epigallocatechin (EGC)
Other: Control — Single oral intake of a flavanol-free, fruit flavored, non-dairy drink.
  Arms: Control

SUMMARY:
The objectives of this study are to i) describe the absorption, distribution, metabolism and excretion (ADME) and pharmacokinetic parameters of selected dietary (poly)phenols in humans; and ii) to compare the ADME and pharmacokinetic parameters of selected dietary (poly)phenols in humans.

DETAILED DESCRIPTION:
Dietary (poly)phenols are a large group of bioactive food constituents that can be classified in flavonoids, stilbenes, lignans and phenolic acids. Flavonoids can be subclassified in different subgroups, including but not limited to flavanols (e.g. (-)-epicatechin, (+)-catechin, procyanidins, EGCG, EGC, etc) and flavones (apigenin and luteolin). Examples of flavanol-containing foods and beverages are apples, chocolate, tea, wine, berries, pomegranate and nuts. Examples of flavone-containing foods and beverages are parsley, celery, and chamomile.

(Poly)phenolic bioactives are actively investigated for their putative beneficial health effects in humans. In this context, understanding the ADME of dietary (poly)phenols is recognized as a key step to gain insight into the nutritional and biomedical relevance of this group of compounds. Understanding the ADME of polyphenols may aid towards i) the identification of metabolites as potential nutritional biomarkers of (poly)phenol consumption, ii) the identification of potential active metabolites mediating the effects observed after (poly)phenol intake, and iii) the design and execution of dietary intervention studies aiming at assess safety and efficacy of (poly)phenols.

Over the last years, significant progress has been made on the description of the ADME of certain (poly)phenols. The investigators recently described the ADME of (-)-epicatechin. However, there is still need to understand the ADME of other polyphenolic bioactives as well as the importance of the role of the gut microbiome in the metabolism of these compounds. In this context, the investigators aim at describing and comparing the ADME of dietary polyphenolic bioactives in humans. To accomplish this, the investigators propose conducting a randomized, double-masked and cross-over dietary intervention study in healthy young adult males. The investigators will evaluate the concentration of polyphenol-derived metabolites in plasma and urine after single acute intakes of polyphenol-containing test materials on 8 different test days.

ELIGIBILITY:
Inclusion Criteria:

* 25-60 years old males
* No prescription medications
* BMI 18.5 - 34.9 kg/m2
* Weight ≥ 110 pounds
* previously consumed cocoa, peanut, parsley, celery and chamomile products with no adverse reactions

Exclusion Criteria:

* Adults unable to consent
* Females
* Prisoners
* Non-English speaking*
* BMI ≥ 35 kg/m2
* Performing vigorous physical activity (i.e. more than 6 MET; metabolic equivalence of task as defined by CDC and ACSM guidelines (http://www.cdc.gov/physicalactivity/everyone/glossary/index.html#vig-intensity; and http://www.cdc.gov/nccdphp/dnpa/physical/pdf/PA_Intensity_table_2_1.pdf ) for more than 3 days a week.
* Dietary allergies including those to nuts, cocoa and chocolate products, parsley, celery and chamomile.
* Active avoidance of either coffee and caffeinated soft drinks
* Under current medical supervision
* A history of cardiovascular disease, stroke, renal, hepatic, or thyroid disease
* History of clinically significant depression, anxiety or other psychiatric condition
* History of Raynaud's disease
* History of difficult blood draws
* Indications of substance or alcohol abuse within the last 3 years
* Current use of herbal, plant or botanical supplements (multi-vitamin/mineral supplements are allowed)
* Blood Pressure > 140/90 mm Hg
* GI tract disorders, previous GI surgery (except appendectomy)
* Self-reported malabsorption (e.g. difficulty digesting or absorbing nutrients from food, potentially leading to bloating, cramping or gas)
* Diarrhea within the last 3 months, or antibiotic intake within the last 3 months
* Vegetarian, Vegan, food faddists, individuals using non-traditional diets, on a weight loss diet or individuals following diets with significant deviations from the average diet
* Metabolic panel and cholesterol results or complete blood counts that are outside of the normal reference range and are considered clinically relevant by the study physician
* Cold, flu, or upper respiratory condition at screening
* Currently participating in a clinical or dietary intervention study

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Changes in the concentration of flavanol metabolites in urine. | Urine collected 12h previous to intervention and up to 24 h after intervention
  Flavanol metabolites include gut microbiome derived metabolites include conjugates of 5-(3',4'-dihydroxyphenyl)-g-valerolactone metabolites and structurally related flavanol conjugated metabolites.
Changes in the concentration of flavanol metabolites in plasma | Plasma collected before (0h) and up to 6h post intervention
  Flavanol metabolites include gut microbiome-derived metabolites like 5-(3',4'-dihydroxyphenyl)-g-valerolactone and structurally related flavanol conjugated metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — UC Davis; Javier I Ottaviani, PhD, Study Director — Mars, Inc.
Locations (1):
- UC Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Only researchers listed in the protocol and approved by the IRB will have access to IPD.

REFERENCES:
- [Background] Schroeter H, Heiss C, Spencer JP, Keen CL, Lupton JR, Schmitz HH. Recommending flavanols and procyanidins for cardiovascular health: current knowledge and future needs. Mol Aspects Med. 2010 Dec;31(6):546-57. doi: 10.1016/j.mam.2010.09.008. Epub 2010 Sep 18. PMID 20854838
- [Background] Ottaviani JI, Momma TY, Kuhnle GK, Keen CL, Schroeter H. Structurally related (-)-epicatechin metabolites in humans: assessment using de novo chemically synthesized authentic standards. Free Radic Biol Med. 2012 Apr 15;52(8):1403-12. doi: 10.1016/j.freeradbiomed.2011.12.010. Epub 2011 Dec 23. PMID 22240152
- [Background] Koster H, Halsema I, Scholtens E, Knippers M, Mulder GJ. Dose-dependent shifts in the sulfation and glucuronidation of phenolic compounds in the rat in vivo and in isolated hepatocytes. The role of saturation of phenolsulfotransferase. Biochem Pharmacol. 1981 Sep 15;30(18):2569-75. doi: 10.1016/0006-2952(81)90584-0. No abstract available. PMID 6946775
- [Background] McCullough ML, Chevaux K, Jackson L, Preston M, Martinez G, Schmitz HH, Coletti C, Campos H, Hollenberg NK. Hypertension, the Kuna, and the epidemiology of flavanols. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S103-9; discussion 119-21. doi: 10.1097/00005344-200606001-00003. PMID 16794446
- [Background] Heiss C, Kleinbongard P, Dejam A, Perre S, Schroeter H, Sies H, Kelm M. Acute consumption of flavanol-rich cocoa and the reversal of endothelial dysfunction in smokers. J Am Coll Cardiol. 2005 Oct 4;46(7):1276-83. doi: 10.1016/j.jacc.2005.06.055. PMID 16198843
- [Background] Del Rio D, Rodriguez-Mateos A, Spencer JP, Tognolini M, Borges G, Crozier A. Dietary (poly)phenolics in human health: structures, bioavailability, and evidence of protective effects against chronic diseases. Antioxid Redox Signal. 2013 May 10;18(14):1818-92. doi: 10.1089/ars.2012.4581. Epub 2012 Aug 27. PMID 22794138
- [Background] Ottaviani JI, Kwik-Uribe C, Keen CL, Schroeter H. Intake of dietary procyanidins does not contribute to the pool of circulating flavanols in humans. Am J Clin Nutr. 2012 Apr;95(4):851-8. doi: 10.3945/ajcn.111.028340. Epub 2012 Feb 29. PMID 22378733